CLINICAL TRIAL: NCT04643795
Title: A Phase I, Open Label, Non-randomized Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Multiple Oral Doses of MGL-3196 in Subjects With Varying Degrees of Hepatic Impairment and Healthy Matched Control Subjects With Normal Hepatic Function
Brief Title: Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Multiple Oral Doses of MGL-3196 in Subjects With Varying Degrees of Hepatic Impairment and Healthy Matched Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-10
Record Dates: First submitted 2020-10-22; First posted 2020-11-25 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Impairment; NASH - Nonalcoholic Steatohepatitis; Cirrhosis, Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 40 mg MGL-3196 Tablet (Experimental): Multiple cohorts (normal, varying hepatic impairment, NASH non-cirrhosis, and NASH cirrhosis) evaluated
  Interventions: Drug: MGL-3196
- 60 mg MGL-3196 Tablet (Experimental): Multiple cohorts (normal, varying hepatic impairment, NASH non-cirrhosis, and NASH cirrhosis) evaluated
  Interventions: Drug: MGL-3196
- 80 mg MGL-3196 Tablet (Experimental): Multiple cohorts (normal, varying hepatic impairment, NASH non-cirrhosis, and NASH cirrhosis) evaluated
  Interventions: Drug: MGL-3196
- 100 mg MGL-3196 Tablet (Experimental): Multiple cohorts (normal, varying hepatic impairment, NASH non-cirrhosis, and NASH cirrhosis) evaluated
  Interventions: Drug: MGL-3196

INTERVENTIONS:
Drug: MGL-3196 — Once daily oral dose for 6 days

SUMMARY:
The purpose of this study is to directly characterize the pharmacokinetic (PK) profiles of MGL-3196 and its major metabolite (MGL-3623) following administration of multiple oral doses (QD x 6 days) in subjects with varying degrees of hepatic impairment (HI) compared to healthy matched control subjects with normal hepatic function, including a subset of NASH subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing and able to sign written informed consent
* Male or female, between 18 and 85 years of age (inclusive)
* BMI between 18 and 45 kg/m2 (inclusive)
* In healthy subjects with normal hepatic function:

  * Considered by the Investigator to be healthy, based on medical and surgical history, physical examination including vital signs, 12-lead ECG, and laboratory test results
  * Match demographically with a subject in the hepatically impaired population according to gender, BMI (±20%), and age (±10 years)
* In subjects with hepatic impairment:

  * Considered by the Investigator to be clinically stable with respect to underlying HI, based on medical and surgical history, physical examination including vital signs, 12-lead ECG, and laboratory test results
* In subjects with NASH:

  * Confirmed diagnosis of NASH suggested by historical data, which include a previous liver biopsy within the last 5 years prior to randomization with evidence of NASH.
  * BMI ≥18 kg/m2

Exclusion Criteria:

* Any clinically significant concomitant disease or condition (including treatment for such conditions) that, in the opinion of the Investigator, could either interfere with the study drug, pose an unacceptable risk to the subject, or compromise interpretation of study data
* Gilbert's syndrome
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of study drug
* eGFR <60 mL/min/1.73 m2 based on Modification of Diet in Renal Disease (MDRD) equation
* Received an investigational drug or device from another study within 30 days (or 5 half-lives, whichever is longer) prior to study drug administration
* In healthy subjects with normal hepatic function:

  * Systolic blood pressure outside the range of 90 to 150 mmHg, diastolic blood pressure outside the range of 40 to 95 mmHg or heart rate outside the range of 40 to 100 beats per minute (bpm)
  * History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months prior to screening
* In subjects with hepatic impairment:

  * Any non-hepatic acute or chronic condition (including, but not limited to, poorly controlled diabetes and encephalopathy Grade ≥3) that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study
  * Acute exacerbation of HI or unstable hepatic function, as determined by the Investigator, 30 days prior to study drug administration
  * Has had a Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure performed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics - Cmax | 16 days
  Cmax after administration
Plasma pharmacokinetics - Tmax | 16 days
  Tmax after administration
Plasma pharmacokinetics - AUC (0-last) | 16 days
  AUC (0-last) after administration
Plasma pharmacokinetics - t1/2 | 16 days
  t1/2 after administration
Effect on the incidence of adverse events | 16 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Madrigal Research Center, Orlando, Florida
  - Madrigal Research Center, Saint Paul, Minnesota
  - Madrigal Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No